CLINICAL TRIAL: NCT00631046
Title: The Importance of Increasing Intake of Essential Fatty Acids During Complementary Feeding on Infant Growth and Body Composition, Intestinal Health, Immune Function and Risk Markers for Later Metabolic Complications.
Brief Title: Essential Fatty Acids During Complementary Feeding
Acronym: EFiON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Axellus (Industry)
Responsible Party: Kim Fleischer Michaelsen, Dr Med Sci, Dept. of Human Nutrition, Rolighedsvej 30, DK-1958 Frederiksberg C, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-A-2007-0088; D203
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Obesity; Growth; Metabolic Syndrome; Cardiovascular Disease
Keywords: n-3 LCPUFA; Fish oil; essential fatty acids; infant growth; obesity; Intestinal microbiota
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Cardiovascular Diseases | interventions — Fish Oils; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fish Oil (Experimental): containing n-3 LCPUFA
  Interventions: Dietary Supplement: Fish Oil
- Sunflower oil (Placebo Comparator): containing n-6 PUFA
  Interventions: Dietary Supplement: Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Daily dosage of 5 ml of fish oils from 9 months +/- 2weeks to 18 months +/- 4 weeks of age
  Arms: Fish Oil
Dietary Supplement: Sunflower Oil — Daily dosage of 5 ml of sunflower oil from 9 months +/- 2weeks to 18 months +/- 4 weeks of age
  Arms: Sunflower oil

SUMMARY:
The objective of this intervention study is to examine the effect of n-3 LCPUFA on growth and body composition, intestinal health and microbiotic composition, immune function and risk markers for later diseases in 9-18 months old infants and toddlers.

ELIGIBILITY:
Inclusion Criteria:

* Singleton infants, 9 mo +/- 2 wk, born >= 37 wk of gestation
* Birth weight >=2500g, a 5-min Apgar score >= 7, birth weight >= 5th percentile for gestational age

Exclusion Criteria:

* Chronic diseases expected to influence growth and dietary intake
* Use of medicine expected to influence growth and dietary intake
* Fish oil supplementation

Ages: 8 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Growth
Body composition
Intestinal microbiota
Blood pressure
Plasma lipid profile
Insulin - glucose
Erythrocyte fatty acid composition
Ex vivo cytokine production
IGF-1 and IGFBP-3
Adipokines
Plasma CRP
Plasma IgE

SECONDARY OUTCOMES:
Glucagon
Metagenome analysis (investigating the enzymatic capacity of the intestines through prokaryotic DNA sequencing)
Iron status (hemoglobin, ferritin)
faecal calprotectin
FADS1 and FADS2 genotypes
Allergy status

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Dr Med Sci, Principal Investigator — Dept. of Human Nutrition, LIFE, Univ. of Copenhagen
Locations (1):
- Dept. of Human Nutrition, Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Lind MV, Martino D, Harslof LB, Kyjovska ZO, Kristensen M, Lauritzen L. Genome-wide identification of mononuclear cell DNA methylation sites potentially affected by fish oil supplementation in young infants: A pilot study. Prostaglandins Leukot Essent Fatty Acids. 2015 Oct;101:1-7. doi: 10.1016/j.plefa.2015.07.003. Epub 2015 Jul 23. PMID 26254087
- [Derived] Harslof LB, Larsen LH, Ritz C, Hellgren LI, Michaelsen KF, Vogel U, Lauritzen L. FADS genotype and diet are important determinants of DHA status: a cross-sectional study in Danish infants. Am J Clin Nutr. 2013 Jun;97(6):1403-10. doi: 10.3945/ajcn.113.058685. Epub 2013 May 1. PMID 23636240
- [Derived] Andersen AD, Molbak L, Michaelsen KF, Lauritzen L. Molecular fingerprints of the human fecal microbiota from 9 to 18 months old and the effect of fish oil supplementation. J Pediatr Gastroenterol Nutr. 2011 Sep;53(3):303-9. doi: 10.1097/MPG.0b013e31821d298f. PMID 21865979